CLINICAL TRIAL: NCT00835393
Title: A Relative Bioavailability Replicated Crossover Study of Pantoprazole Sodium 40 mg DR Tablets Under Non-Fasting Conditions.
Brief Title: Pantoprazole Sodium 40 mg DR Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B036582
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pantoprazole Sodium 40 mg delayed-release tablets
- 2 (Active Comparator)
  Interventions: Drug: PROTONIX® 40 mg delayed-release tablets.

INTERVENTIONS:
Drug: Pantoprazole Sodium 40 mg delayed-release tablets — 1 x 40 mg
  Arms: 1
Drug: PROTONIX® 40 mg delayed-release tablets. — 1 x 40 mg
  Arms: 2

SUMMARY:
The Objective of this study is to compare the relative bioavailability of pantoprazole sodium 40 mg delayed-released tablets (manufactured by TEVA Pharmaceutical Industries,Ltd. and distributed by TEVA Pharmaceuticals USA)with that of PROTONIX® 40mg delayed-released tablets (Wyeth- Ayerst) in Healthy, adult, non-smoking subjects under non- fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be non-smokers at least 18 years of age. Subjects will have a BMI (Body Mass Index) of 30 or less.

Exclusion Criteria:

* Subjects with a significant recent history of chronic alcohol consumption (past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular, disease, tuberculosis, epilepsy, asthma (past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result not to be significant.
* Subjects who have a history of allergic responses to the class of drug being tested will be excluded from the study.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each dosing period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/ot plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives anytime during the 180 days prior to study dosing or oral hormonal contraceptives with in 14 days of dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be with drawn from the study.
* Subjects who do not tolerate venipuncture will not be allowed to participate.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Steven Herrmann, M.D.; Ph.D, Principal Investigator — Cetero Research, San Antonio
Locations (2):
- United States (2):
  - Gateway Medical Research, Inc., Saint Charles, Missouri
  - Bioassay Laboratory, Inc., Houston, Texas